CLINICAL TRIAL: NCT05429866
Title: Immunological Variables Associated to ICI Toxicity in Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Principal Investigator, Mireille Langouo Fontsa, Principal investigator, Jules Bordet Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IJB-IRAES-2020
Record Dates: First submitted 2022-04-24; First posted 2022-06-23 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Melanoma; Non Small Cell Lung Cancer; Non-melanoma Skin Cancer; Gastrointestinal Cancer; Head and Neck Cancer; Renal Cell Carcinoma; Small Cell Lung Cancer; Mesothelioma, Malignant; Bladder Cancer; Merkel Cell Carcinoma; Hepatocellular Carcinoma; MSI-H Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung; Gastrointestinal Neoplasms; Head and Neck Neoplasms; Carcinoma, Renal Cell; Small Cell Lung Carcinoma; Mesothelioma, Malignant; Urinary Bladder Neoplasms; Carcinoma, Merkel Cell; Carcinoma, Hepatocellular | interventions — Immune Checkpoint Inhibitors; Nivolumab; atezolizumab; avelumab; durvalumab; cemiplimab

STUDY DESIGN:
Intervention Model Description: This is a monocentric, prospective, pilot study that will enrol 435 subjects with solid tumours that are treated with immune checkpoint inhibitor(s) (ICI) alone or in combination with chemotherapy or targeted therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Checkpoint Blockade, Immune — Immune checkpoint blockade drugs target the immune system by blocking control pathways regulating anti-tumor immunity and thereby reinvigorate their activities against cancer.
  Other Names: Ipililumab; Nivolumab; Pembrozilumab; atezolizumab; avelumab; durvalumab; Cemiplimab

SUMMARY:
This is a monocentric, prospective, pilot study that will enrol 435 subjects with solid tumours that are treated with immune checkpoint inhibitor(s) (ICI) alone or in combination with chemotherapy or targeted therapy.

For enrolled subjects, clinical and laboratory evaluations will be performed and reported at different time points:

* Early (4-6 weeks after treatment start)
* Midtime (8-11 weeks after treatment start)
* Late (13-18 weeks after treatment start)
* At the occurrence of immune-related adverse events (irAEs), clinical and laboratory evaluation will be performed at two principal time points:

  * For the 1st time of any grade 1 or 2 irAE if the subject developed it.
  * For the 1st time of any grade 3 or 4 irAE if the subject developed it.

DETAILED DESCRIPTION:
Advances in treating patients with immunotherapy has dramatically changed cancer morbidity and mortality. Immune checkpoint inhibitors (ICI), alone or combined with other drugs, are currently used both as standard of care or in experimental settings for various cancers. Currently, ICI treatment induces objective clinical responses in 20-40% of patients, which varies by tumour type. A significant risk of immune-related adverse events (irAE) is also associated with ICI treatment, including the onset of autoimmune diseases. While the incidence of irAE is highly variable and influenced by many factors, phase I and II trials reported rates from 10% to 80% for any grade irAE while an irAE of grade 3 or higher was observed in 2.5% to 18% of subjects. Despite the fact that older adults represent the growing majority of patients diagnosed with cancer, the efficacy and toxicity of ICI in older patients, alone or in combination with other agents, remains controversial. Presently, the specific immune mechanism(s) driving irAE are unknown and biomarkers that predict their onset, particularly high-grade irAE, are urgently needed. The identification of predictive clinical, laboratory and immunological biomarkers (blood and tissue) for toxicity will more accurately identify and quantify patients who are at risk for ICI therapy. Then, this will possibly allow better irAE management.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥ 18 years old
* 2) ECOG performance status ≤ 1
* 3) Must have histologically or cytologically confirmed solid tumour, eligible for treatment with ICI as standard-of-care alone or in combination with another ICI (cohort 1), ICI with chemotherapy (cohort 2), or ICI with targeted therapy (cohort 3) with no restrictions on number of prior systemic therapies
* 4) All prior anti-cancer treatment-related toxicities (except alopecia) must be ≤ Grade 1 according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 at the time of enrolment
* 5) Serum pregnancy test (for subjects of childbearing potential) negative within 15 days prior to study medications administration.
* 6) Women of childbearing potential must agree to use one highly effective method of contraception prior study entry, during the course of the study and at least 7 months after the last administration of study treatments.
* 7) Men with childbearing potential partner must agree to use condom during the course of this study and for at least 6 months after the last administration of the study treatments.
* 8) Completion of all necessary screening procedures within 14 days prior to enrolment.
* 9) Signed Informed Consent form (ICF) obtained prior to any study related procedure.

Exclusion Criteria:

* Subjects meeting one of the following criteria are not eligible for this study:

  1. Subject with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study.
  2. Participation in another clinical trial.
  3. Pregnant and/or lactating women.
  4. Subjects already receiving ICI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Modification(s) in the immune blood markers of treated subjects on treatment. | Assessment: between week 4 and 6 after the first dose of the treatment
  Modification(s) in the immune blood markers including cytokines, immune cells and serum autoantibody level of treated subjects.
Modification(s) in the immune blood markers of treated subjects on treatment. | Assessment: between week 8 and 11 after the first dose of the treatment
  Modification(s) in the immune blood markers including cytokines, immune cells and serum autoantibody level of treated subjects.
Modification(s) in the immune blood markers of treated subjects on treatment. | Assessment: between week 13-18 after the first dose of the treatment
  Modification(s) in the immune blood markers including cytokines, immune cells and serum autoantibody level of treated subjects.
Modification(s) in the immune blood markers of treated subjects on treatment at the occurence of any grade 1 or 2 irAE. | Assessment: Day1 after diagnostic of any grade 1 or 2 irAE
  Safety will be assessed and graded by the investigator(s) by using the adverse events reported during the study in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Modification(s) in the immune blood markers of treated subjects on treatment at the occurence of any grade 3 or 4 irAE. | Assessment: Day one after diagnostic of any grade 3 or 4 irAE
  Safety will be assessed and graded by the investigator(s) by using the adverse events reported during the study in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Anderlecht, Belgium

IPD SHARING:
Plan to Share IPD: No